CLINICAL TRIAL: NCT02736721
Title: Multicenter Open Label Expanded Access-Program of Pegylated Interferon Alfa-2a (Pegasys) in Patients With Chronic Myelogenous Leukemia (CML)
Brief Title: Expanded Access Study With Peginterferon Alfa-2a (Pegasys) in Participants With Chronic Myelogenous Leukemia (CML)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML17395
Record Dates: First submitted 2016-04-08; First posted 2016-04-13 (Estimated); Results first posted 2016-08-05 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-05

CONDITIONS: Myelogenous Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — peginterferon alfa-2a

ARMS (1):
- Peginterferon alfa-2a (Experimental): Participants will receive peginterferon alfa-2a subcutaneously in doses between 90 and 450 microgram (mcg) once weekly until medically indicated as judged by the treating investigator.
  Interventions: Drug: Peginterferon alfa-2a

INTERVENTIONS:
Drug: Peginterferon alfa-2a — Peginterferon alfa-2a in doses between 90 and 450 mcg will be administered subcutaneously once weekly until medically indicated as judged by the treating investigator.
  Other Names: Pegasys

SUMMARY:
This study will evaluate the efficacy, safety and tolerability of long-term use of peginterferon alfa-2a in participants with CML who have previously participated in peginterferon alfa-2a study ML16544 (NCT number not available), NO16006 (NCT number not available) or ML17228 (NCT number not available) and treating physician has decided to continue treatment with peginterferon alfa-2a within the frame of another clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with CML
* Previous participation in studies: ML16544, NO16006 or ML17228; for which the treating physician recommends a continuation of the study drug according to defined minimal criteria

Exclusion Criteria:

* Major protocol violator in the participated study prior to participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2003-09; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (5):
- Germany (5):
  - Freiburg im Breisgau
  - Mainz
  - Mannheim
  - Marburg
  - Tübingen

RESULTS

PARTICIPANT FLOW:
Groups:
- Peginterferon Alfa-2a: Participants who have previously participated in study ML16544 (NCT number not available), NO16006 (NCT number not available) or ML17228 (NCT number not available) and deemed to be a responder, received peginterferon alfa-2a subcutaneously in doses between 90 and 450 microgram (mcg) once weekly until medically indicated as judged by the treating investigator. Maximum treatment duration was approximately up to 7 years.
Period: Overall Study
Arm/Group | Peginterferon Alfa-2a
Started | 41
Completed | 25
Not Completed | 16
Not completed — Adverse Event | 8
Not completed — Lost to Follow-up | 3
Not completed — Other | 5

BASELINE CHARACTERISTICS:
Population: Analysis population included all enrolled participants.
Groups:
- Peginterferon Alfa-2a: Participants who have previously participated in study ML16544, NO16006, or ML17228 and deemed to be a responder, received peginterferon alfa-2a subcutaneously in doses between 90 and 450 mcg once weekly until medically indicated as judged by the treating investigator. Maximum treatment duration was approximately up to 7 years.
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Hematologic Response
Description: Hematologic response was considered to be achieved if participants met all of the following criteria: normalization of white blood cells count to less than (<) 10*10^9 per liter (/L) with normal differentiation, normalization of platelet count at <450*10^9/L, and disappearance of all signs and symptoms of the disease. This response had to be confirmed at least 4 weeks after the first measure and beyond that.
Time Frame: Up to approximately 7 years
Population: Analysis population included all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 41
participants | 40

2. Primary Outcome: Time to Loss of Previous Hematologic Response
Description: Time to loss of previous hematologic response was defined as the interval between the first day of treatment in the study and the first day of loss of previous hematologic response during elapsed time of study. Hematologic response was considered to be achieved if participants met all of the following criteria: normalization of white blood cells count to <10*10^9/L with normal differentiation, normalization of platelet count at <450*10^9/L, and disappearance of all signs and symptoms of the disease. This response had to be confirmed at least 4 weeks after the first measure and beyond that.
Time Frame: Up to approximately 7 years
Population: Analysis population included all enrolled participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 41
months | NA [NA to NA] — The median and corresponding 95% confidence interval (CI) data was not estimable because only 1 participant, out of total 41 participants, lost previous hematological response.

3. Primary Outcome: Number of Participants With Major Cytogenetic Response (CyR)
Description: CyR was based on the prevalence of Philadelphia chromosome-positive (Ph+) bone marrow cells in metaphase determined from reverse transcriptase polymerase chain reaction (RT-PCR). Major cytogenetic response was categorized as either complete cytogenetic response (CCyR) or partial cytogenetic response (PCyR). CCyR was achieved when there was absence of detectable Ph+ bone marrow cells and PCyR was achieved when 1 to 34 percent (%) of bone marrow cells were Ph+.
Time Frame: Up to approximately 7 years
Population: Analysis population included all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 41
participants | 40

4. Primary Outcome: Time to Loss of Previous CyR
Description: Time to loss of previous CyR was defined as the interval between the first day of treatment in the study and the first day of loss of previous CyR. CyR is based on the prevalence of Ph+ bone marrow cells in metaphase. Major CyR was categorized as either CCyR or PCyR. CCyR was achieved when there was absence of detectable Ph+ bone marrow cells and PCyR was achieved when 1 to 34% of bone marrow cells were Ph+.
Time Frame: Up to approximately 7 years
Population: Analysis population included all enrolled participants.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 41
years | NA [NA to NA] — The median and corresponding 95% CI data was not estimable because only 1 participant, out of total 41 participants, lost previous CyR.

5. Primary Outcome: Number of Participants With Molecular Response (MR)
Description: MR was assessed using breakpoint cluster region - Abelson (BCR-ABL) proto-oncogene transcript levels measured by RT-PCR from peripheral blood. Number of participants with BCR-ABL/ABL ratio less than or equal to 10 (%) was reported.
Time Frame: Up to approximately 7 years
Population: Analysis population included all enrolled participants.
Measure: Number; unit: participants
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 41
participants | 38

6. Primary Outcome: Time to Loss of Previous MR
Description: Time to loss of previous MR was defined as the interval between the first day of treatment in the study and the first day of loss of previous MR. MR was assessed using BCR-ABL transcript levels measured by RT-PCR from peripheral blood.
Time Frame: Up to approximately 7 years
Population: Analysis population included all enrolled participants.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Peginterferon Alfa-2a
Number analyzed (Participants) | 41
years | NA [NA to NA] — The median and corresponding 95% CI data was not estimable because limited number of participants lost previous MR.

ADVERSE EVENTS:
Time Frame: Up to approximately 7 years
Description: Analysis population included all enrolled participants.
Arm/Group | Peginterferon Alfa-2a
Serious Adverse Events (participants affected / at risk) | 13/41
Other Adverse Events (participants affected / at risk) | 35/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a (N=41)
Atrial fibrillation (Cardiac disorders) | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Depression (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Colostomy (Surgical and medical procedures) | 1
Finger amputation (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a (N=41)
Neutropenia (Blood and lymphatic system disorders) | 4
Leukopenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Nausea (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 5
Influenza like illness (General disorders) | 5
Pyrexia (General disorders) | 4
Oedema (General disorders) | 3
Bronchitis (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 4
Cystitis (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Depression (Psychiatric disorders) | 7
Erythema (Skin and subcutaneous tissue disorders) | 5
Night sweats (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.